CLINICAL TRIAL: NCT03889964
Title: Reduced Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease -Relevance of Cardiovascular Comorbidities
Brief Title: Exercise Capacity in COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: 17-033
Record Dates: First submitted 2019-03-11; First posted 2019-03-26 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: cardiopulmonary exercise testing; cardiovascular comorbidities; cardiopulmonary interaction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of 20 ml of peripheral blood Clinical routine such as NTproBNP, renal function, thyroid function, blood count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with stable COPD
  Interventions: Other: Measurement of lung function, electrocardiography, echocardiography and cardiopulmonary exercise testing

INTERVENTIONS:
Other: Measurement of lung function, electrocardiography, echocardiography and cardiopulmonary exercise testing — Measurement of lung function, electrocardiography, echocardiography and cardiopulmonary exercise testing

SUMMARY:
In this study, cardiopulmonary exercise will be assessed to characterize the relevance of severity of COPD and coexisting cardiovascular comorbidities for exercise capacity.

DETAILED DESCRIPTION:
In patients with chronic obstructive pulmonary disease (COPD) the interpretation of dyspnoea also needs to consider coexisting cardiovascular disease. Cardiopulmonary exercise testing (CPET) is used to characterize pulmonary and cardiac function and limitations during exercise. The investigators hypothesise that cardiopulmonary exercise is reduced in COPD patients with coexisting cardiovascular disease as well as in more symptomatic patients and in patients with frequent exacerbations. For this purpose, 100 patients with with stable COPD are characterized by clinical characteristics, laboratory tests, lung function, electrocardiography, echocardiography and cardiopulmonary exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* patients with stable chronic obstructive pulmonary disease, exacerbated or stable
* 40-80 years
* sinus rhythm
* informed written consent

Exclusion Criteria:

* Inability to give written consent
* acute myocardial infarction with ST-segment elevations in last 30 days
* severe acute or chronic renal dysfunction
* severe heart failure-
* atrial fibrillation
* severe valve disease
* severe hypoxemia
* long term oxygen therapy or non invasive ventilation

Ages: 40 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Patients with stabile chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of oxygen uptake during cardiopulmonary exercise testing (% predicted) | Baseline

SECONDARY OUTCOMES:
measurement of dyspnoea quantified by the COPD assessment test as well as the modified Medical Research Council Scale | Baseline
  For the assessment of the symptoms of the study group and its relation to exercise capacity dyspnoea is assessed by accepted questionnaires typically used for COPD patients at baseline
Measurement of FEV1 | Baseline
Measurement the capillary pO2 in mmHg and capillary pCO2 at baseline | Baseline
  The blood gases pO2 and pCO2 are taken from the hyperaemic ear lobe to characterize the gas exchange during cardiopulmonary exercise which is a routine procedure
N-terminal pro brain natriuretic peptid (NTproBNP) in ng/L from peripheral venous blood at baseline | Baseline
  NTproBNP is analysed from peripheral venous blood to characterize potential heart failure and its relation to exercise capacity of the study subjects
Measurement of Maximum wattage during cardiopulmonary exercise testing | Baseline
Measurement of Breathing reserve during cardiopulmonary exercise testing | Baseline
  BThe breathing reserve in % is assessed at the end of the cardiopulmonary exercise testing to characterize a ventilatory limitation of the exercise test. It is calculated as percent from the minute ventilation in relation to the maximum mandatory ventilation. The measurement is a routine measurement during cardiopulmonary exercise testing.
Measurement of Oxygen pulse during cardiopulmonary exercise testing | Baseline
Presence of cardiovascular comorbidities | Baseline
  For the cardiopulmonary characterization clinical characteristics, lung function, blood gases, laboratory investigation, ECG and echocardiography were used in addition to cardiopulmonary exercise testing.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Düsseldorf, Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided